CLINICAL TRIAL: NCT00682448
Title: Metformin to Prevent the Metabolic Complications of Olanzapine
Brief Title: Metformin for the Prevention of the Metabolic Side-effects of Zyprexa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jeffrey Rado, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06122201
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Metabolic Complications
Keywords: Olanzapine; Zyprexa; Weight Gain; Antipsychotics; Metformin; Glucophage; Bipolar Disorder; Schizophrenia; Depression; Diabetes; Side effects; Metabolic complications; Prevention; Treatment; Metabolic side effects of olanzapine
MeSH Terms: conditions — Weight Gain; Bipolar Disorder; Schizophrenia; Depression; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Olanzapine plus metformin: olanzapine plus metformin 500 mg titrated up to but no greater than 2,000 mg based upon fasting blood glucose during study visits over six months.
  Interventions: Drug: Metformin
- 2 (Placebo Comparator): Olanzapine plus Drug: Placebo. Subjects will remain on olanzapine plus placebo for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Drug: Metformin 500 mg po daily titrated up to but no greater than 2000 mg based upon fasting blood glucose during study visits over six months.
  Other Names: Glucophage; Fortamet; Riomet; Glumetza; Diabex; Diaformin
  Arms: 1
Drug: Placebo — Drug: Placebo. Subjects will remain on placebo for 6 months.
  Arms: 2

SUMMARY:
We hypothesize that metformin co-administered with olanzapine will be well tolerated and associated with significantly less insulin resistance, weight gain and dyslipidemia as compared to olanzapine plus placebo.

DETAILED DESCRIPTION:
Increased risk of metabolic complications with olanzapine therapy, relative to other antipsychotics, may lead clinicians to avoid its use, despite evidence of greater efficacy. These problems may also pose a therapeutic dilemma for patients who respond well to olanzapine. Metabolic complications negatively impact on morbidity and mortality, impair quality of life and increase illness relapse secondary to medication non-compliance. Thus far, no pharmacologic agent co-administered with olanzapine has proven effective at preventing these untoward effects. The present study proposes to examine the efficacy and safety of metformin to attenuate the metabolic side effects associated with olanzapine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of: Schizophrenia, Schizoaffective Disorder, Bipolar I or II or major depression with psychotic features who will be started on or who have just started taking Olanzapine (Zyprexa).

Exclusion Criteria:

* Patients with either a history of diabetes mellitus or a baseline FBG>126 or two random blood sugars of > 200 or during a OGTT glucose level of > 200 two hours after a glucose load of 50 grams. (All American Diabetes Association criteria for diabetes mellitus).
* Baseline liver function tests (SGOT, SGPT, AP) greater than 3X normal.
* Chronic alcoholism
* MDRD less than 60 ml/1.73 m2. Modification of Diet in Renal Disease (MDRD) Equation estimates the glomerular filtration rate as a measure of kidney function. This equation takes into account the plasma creatinine, age, race and gender, and is a more accurate estimation of glomerular filtration rate than serum creatinine alone.
* Patients with unstable medical problems, including cardiovascular instability or significant congestive heart failure (as determined by study investigators).
* Prolonged QTc greater than 430 ms on baseline EKG.
* History of lactic acidosis.
* History of hypoglycemia.
* Current treatment with metformin or other antidiabetic agents.
* Treatment with any antihyperlipidemic medication within 3 months of randomization.
* Treatment with olanzapine or clozapine within 3 months of randomization.
* Concurrent treatment with ziprasidone, risperidone, quetiapine or aripiprazole or any other neuroleptic medication.
* Concurrent use of OTC chromium, gymnema or cimetidine will be prohibited. Patient may discontinue these medications up to one day prior to randomization.
* Current treatment with corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Rado, M.D., Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Olanzapine plus metformin: olanzapine plus metformin 500 mg titrated up to but no greater than 2,000 mg based upon fasting blood glucose during study visits over six months.
  Metformin: Drug: Metformin 500 mg po daily titrated up to but no greater than 2000 mg based upon fasting blood glucose during study visits over six months.
- Placebo: Olanzapine plus Drug: Placebo. Subjects will remain on olanzapine plus placebo for 6 months.
  Placebo: Drug: Placebo. Subjects will remain on placebo for 6 months.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 12 | 13
Completed | 7 | 7
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Men and women age 18 and over with schizophrenia, schizoaffective disorder, bipolar disorder or Major depression with psychotic features.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.12) | 39.08 (8.62) | 36.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 3 | 12
  African American | 4 | 8 | 12
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 27
weight [Mean (Standard Deviation); unit: kilogram] | 84.51 (16.56) | 95.59 (34.44) | 90.33 (27.39)

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain
Description: Change from Baseline in weight
Time Frame: Baseline and 6 months
Population: intent to treat using last observation carried forward. Only subjects with one observation post-baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 13
kilogram | 2.54 (2.35) | 5.88 (5.23)

2. Secondary Outcome: Hemoglobin A1C
Description: change from baseline in hemoglobin AIC
Time Frame: Baseline and 6 months
Population: total of 18 participants reflects the number of participants with available data at 6 months.
Measure: Mean (Standard Deviation); unit: % HbAIC
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 10 | 8
% HbAIC | 0.05 (0.28) | 0.1 (0.26)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/13
Other Adverse Events (participants affected / at risk) | 3/12 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=12) | Placebo (N=13)
suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) — suicidal ideation
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=12) | Placebo (N=13)
sedation (Psychiatric disorders) | 3 (3) | 3 (3) — sedation
Dry mouth (Endocrine disorders) | 3 (3) | 5 (5) — dry mouth
stomach upset (Gastrointestinal disorders) | 3 (3) | 6 (6) — stomach complaints including nausea, constipation, diarrhea
headache (Nervous system disorders) | 3 (3) | 1 (1) — headache
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — low blood sugar

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No